CLINICAL TRIAL: NCT03810716
Title: Promotion of Family Planning Methods Through an Interactive Platform Offered in Growth and Development Control Services
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Peruana Cayetano Heredia (Other)
Responsible Party: Principal Investigator, Suzzane Minaya Romero, Principal Investigator, Universidad Peruana Cayetano Heredia
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SIDISI: 102347
Record Dates: First submitted 2018-10-08; First posted 2019-01-22 (Actual); Last update posted 2019-01-22 (Actual); Status verified 2019-01

CONDITIONS: Women
Keywords: interactive platform; family planning; contraception

STUDY DESIGN:
Intervention Model Description: Quasi - experimental study design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interactive Platform (Experimental): Tha participants in this group will see the interactive platform and answer a survey before and after the intervention. Their clinical health records will be checked one month ago.
  Interventions: Device: Interactive Platform
- Control (No Intervention): The participants in this group will answer the survey. Their clinical health records will be checked one month ago.

INTERVENTIONS:
Device: Interactive Platform — The participants will see the interactive platform.
  Arms: Interactive Platform

SUMMARY:
Family planning and the use of contraceptive methods are of the main strategies to reduce maternal and perinatal morbidity and mortality, because they can prevent unplanned pregnancies, teenage pregnancies and abortions in dangerous conditions. It is also a tool that contributes to development as it improves children's health, improves access to early childhood education, empowers women and contributes to reducing poverty as it improves economic conditions.

Currently the use of modern contraceptive methods has increased worldwide, in Latin America and the Caribbean the use of modern contraceptive methods has remained at 66.07% from 2008 to 2015. However, the number of women who do not want to get pregnant and that do not use a contraceptive method is still high - 214 million women of childbearing age in developed countries.

In our country according to the ENDES 2016 survey, the number of women who used a contraceptive method decreased by 0.7 percent compared to 2012, of which 54.3 percent used some modern contraceptive method and 21.9 percent some method traditional.

The unmet demand for family planning in 2016 was 6.0%, affecting mainly women from the lowest poverty quintile (7.4%) and those living in rural areas (6.8%).

Of the women who were surveyed and did not use a contraceptive method, 80.6% did not talk about family planning either at home or in a health facility in the last 12 months. Only 16.3% of non-users were women who attended a health facility and received information on family planning.

Through this study the investigators propose the design and evaluation of an interactive platform to promote modern contraceptive methods.

DETAILED DESCRIPTION:
Sample Size: Sample size of 176 participants (interventional group=88, control group=88), it is possible to detect minimum differences of 5% to 20%.

Statistical analysis plan: The data collected will be entered into a database in Microsoft Excel, to be analyzed by the Epi Info statistical program. The qualitative variables will be analyzed by frequencies and percentages, the quantitative variables by relative risk.

ELIGIBILITY:
Inclusion Criteria:

* Mothers of children who attend the service of growth and development who are of legal age
* Women who do not currently use some modern contraceptive method
* Women whose partners have not received voluntary surgical contraception

Exclusion Criteria:

* Teen mothers
* Illiterate women
* Women who currently do not have a partner
* Women who are currently gestating

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 176 (Actual)
Dates: Start 2018-10-29 (Actual); Primary Completion 2018-12-27 (Actual); Study Completion 2018-12-27 (Actual)

PRIMARY OUTCOMES:
Percentage of mothers who attend the family planning service | one month
  Percentage of women who assist to family planning service after the intervention

SECONDARY OUTCOMES:
Percentage of mothers who initiate a contraceptive method | one month after the intervention
  Percentage of mothers who initiate a contraceptive method after the intervention
Satisfaction of the users about the interactive platform | immediately after the intervention
  The participants will answer a survey to rate usability after the intervention. This survey is a likert survey.

CONTACTS AND LOCATIONS:
Overall Officials: Suzzane S Minaya Romero, BSc, Principal Investigator
Locations (2):
- Peru (2):
  - Cueto Fernandini, Lima, Los Olivos
  - Los Olivos, Lima, Los Olivos

IPD SHARING:
Plan to Share IPD: No
There is no plan description. No applicable.

REFERENCES:
- [Result] Sheoran B, Braun RA, Gaarde JP, Levine DK. The hookup: collaborative evaluation of a youth sexual health program using text messaging technology. JMIR Mhealth Uhealth. 2014 Nov 3;2(4):e51. doi: 10.2196/mhealth.3583. PMID 25367444
- [Result] Mishra N, Panda M, Pyne S, Srinivas N, Pati S, Pati S. Barriers and enablers to adoption of intrauterine device as a contraceptive method: A multi-stakeholder perspective. J Family Med Prim Care. 2017 Jul-Sep;6(3):616-621. doi: 10.4103/2249-4863.222028. PMID 29417019
- [Result] Ngum Chi Watts MC, Liamputtong P, Carolan M. Contraception knowledge and attitudes: truths and myths among African Australian teenage mothers in Greater Melbourne, Australia. J Clin Nurs. 2014 Aug;23(15-16):2131-41. doi: 10.1111/jocn.12335. Epub 2013 Sep 13. PMID 24028778
- [Result] Ewerling F, Victora CG, Raj A, Coll CVN, Hellwig F, Barros AJD. Demand for family planning satisfied with modern methods among sexually active women in low- and middle-income countries: who is lagging behind? Reprod Health. 2018 Mar 6;15(1):42. doi: 10.1186/s12978-018-0483-x. PMID 29510682
- See also: LA PLANIFICACIÓN FAMILIAR COMO HERRAMIENTA BÁSICA PARA EL DESARROLLO FAMILY PLANNING AS A BASIC TOOL FOR DEVELOPMENT — http://www.scielo.org.pe/pdf/rins/v30n3/a16v30n3.pdf